CLINICAL TRIAL: NCT00148863
Title: Pilot Study on Interferon Gamma in Association With Peg-Interferon Alpha 2a and Ribavirin Among Patients With a Chronic Hepatitis C and Non Responders to the Association of Peg-Interferon Alpha 2b or 2a and Ribavirin ANRS HC16 Gammatri
Brief Title: Interferon Gamma With Peg-Interferon Alpha 2a and Ribavirin in Non Responders Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: InterMune (Industry); Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-005033-19; ANRS HC16 Gammatri
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2007-08-30 (Estimated); Status verified 2007-08

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Interferon Alfa-2a; Ribavirin; Interferon-gamma, Recombinant
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Pharmaceutical Preparations; Ribavirin; Interferon-gamma

INTERVENTIONS:
Drug: Peg-interferon alpha 2a (drug)
Drug: Ribavirin (drug)
Drug: Interferon gamma (drug)

SUMMARY:
Viral hepatitis C is treated with peg-interferon alpha 2a/2b and ribavirin. There is no treatment recommended for non responders patients. This study will evaluate the efficacy, after a second treatment with peg-interferon alpha 2a and ribavirin for 12 Weeks of the addition of interferon gamma in non responders patients

DETAILED DESCRIPTION:
Viral hepatitis C is treated with peg-interferon alpha 2a/2b and ribavirin for 24 Weeks. In many patients, there is no efficacy of this treatment on hepatitis C, and there is no treatment recommended for them. Interferon gamma has anti-infectious and anti-fibrosis activity. This study will evaluate the effect, after a second treatment with peg-interferon alpha 2a and ribavirin for 12 Weeks, of the addition of interferon gamma in non responders patients. 65 patients will be included in order to include 27 patients who are non responders after 12 weeks of a second treatment and are eligible to receive interferon gamma. Patients will then receive peg-interferon alpha 2a (180 micro g once a week, by injection), ribavirin (1,000 to 1,200 mg per day, according to weight) and interferon gamma (100 micro g thrice a week, by injection) during 8 months

ELIGIBILITY:
Inclusion Criteria:

* Positive anti-HCV antibodies
* Positive HCV RNA (quantitative method)
* Previous treatment with Peg-interferon alpha 2b 1.0 to 1.5 micro g/kg (during at least 12 weeks) with ribavirin (at least 800 mg/day during at least 12 weeks),stopped since at least 3 months
* Without lower dosage during previous treatment
* Non responder to the previous treatment with Peg-interferon alpha 2b and ribavirin, with detectable HCV RNA at W24 or decrease of less than 2 log10 copies/ml at W12 or decrease greater than 2 log10 but detectable HCV RNA
* Metavir over F2 on the most recent biopsy
* ALT increase over normal value twice during last 6 months

Exclusion Criteria:

* HIV infection
* Psychiatric pathology
* Alcool consummation
* Cirrhosis
* Pregnancy or plan of pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2004-06; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Virological response as defined by an HCV RNA measure non detectable at W28 with qualitative PCR (centralized measure)

SECONDARY OUTCOMES:
Virological response at W72
Biochemical response at W72 (ALT below normal value)
Quality of life
Immunologic response (CD4 and CD8 HCV specific)
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Patrice Couzigou, MD, PhD, Principal Investigator — Hôpital du Haut-Lévêque, Pessac, France; Geneviève Chêne, MD, PhD, Study Director — INSERM U593, Bordeaux, France
Locations (2):
- France (2):
  - Hopital Haut Leveque Service d'Hepato-Gastro-Enterologie, Pessac
  - Hôpital du Haut-Levêque, Pessac

REFERENCES:
- [Derived] Couzigou P, Perusat S, Bourliere M, Trimoulet P, Poynard T, Leroy V, Marcellin P, Foucher J, Bronowicki JP, Chene G; ANRS HC16 GAMMATRI Trial Group. Interferon-gamma with peginterferon alpha-2a and ribavirin in nonresponder patients with chronic hepatitis C (ANRS HC16 GAMMATRI). J Gastroenterol Hepatol. 2013 Feb;28(2):329-34. doi: 10.1111/jgh.12060. PMID 23190183